CLINICAL TRIAL: NCT06842888
Title: Comparing Mirror Therapy Rehabilitation Device to Conventional Mirror Therapy
Acronym: MiraPi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000039425
Record Dates: First submitted 2025-02-18; First posted 2025-02-24 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Stroke; Pain; Impaired Motor Function
MeSH Terms: conditions — Stroke; Pain | interventions — Mirror Movement Therapy

STUDY DESIGN:
Intervention Model Description: Inpatients undergoing inpatient rehabilitation in the IRU (inpatient rehabilitation unit) at the Yale New Haven Hospital Rehabilitation and Wellness Center
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional Therapy Group (Active Comparator): Participants in this group with train using Mirror Therapy (MT), the current standard of care, performing it on the affected arm for 15 minutes daily, 3 days per week until their discharge from clinic (approximately 2-3 weeks).
  Interventions: Behavioral: Mirror Therapy
- Miraπ Group (Experimental): Participants in this group will train with the Miraπ device, performing it on the affected arm for 15 minutes daily, 3 days per week until their discharge from clinic (approximately 2-3 weeks).
  Interventions: Device: Miraπ

INTERVENTIONS:
Device: Miraπ — This device has tiny sensors that measure the movement of the healthy fingers and tiny motors that move the affected fingers of the patient.
  The device is connected to a specially designed finger mechanism that moves the affected fingers of the patient. This opening mechanism is designed in a way that it prevents the fingers from being forced into any hurting position. If the patient moves the healthy fingers during training, also the fingers of the affected hand are moved by the device at the same time. This creates the effect of mirror therapy for the brain as the patient can see both hands moving.
  Arms: Miraπ Group
Behavioral: Mirror Therapy — Current standard of care using MT.
  Arms: Conventional Therapy Group

SUMMARY:
This is a randomized controlled trial which will compare conventional mirror therapy with mirror therapy using the Miraπ device which physically moves a patient's affected limb.

This study will use two parallel groups: (1) receiving conventional mirror therapy as a part of the standard of care as conducted by the participant's clinical care team and (2) receiving mirror therapy with the Miraπ device as conducted by study personnel with the oversight of the participant's clinical care team.

ELIGIBILITY:
Inclusion Criteria:

* Participants currently accepted and cleared for rehabilitation in the inpatient rehabilitation unit by the rehabilitation medical director.
* Participants with paralysis or motor function problems of only one hand.
* Participants need mirror therapy because of their health condition.
* Participants' rehabilitation physician determined that mirror therapy would be appropriate for standard of care.
* Participants are able to memorize easy tasks, and able to follow instructions e.g., moving the healthy fingers.

Exclusion Criteria:

* Participants who are not cleared physically or medically to participate in standard acute inpatient rehabilitation therapies by the rehabilitation medical director
* Participants who are not able to memorize easy tasks, e.g., moving the healthy fingers.
* Participants with spasticity of the affected hand (as assed by the occupational therapist)
* Minors
* Vulnerable populations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2025-03-31 (Actual); Primary Completion 2025-08-19 (Actual); Study Completion 2025-08-19 (Actual)

PRIMARY OUTCOMES:
Change in Jebsen-Taylor Hand Function Test score | At baseline and at discharge (approximately 2-3 weeks after baseline)
  Percentage score, which determines how well a participant can do motor tasks for range of motion, strength, and tasks of activities of daily life. Participants have up to 120 seconds to complete tasks. Lower scores indicate less impairment.
McGill Pain Questionnaire (MPQ) | At baseline and at discharge (approximately 2-3 weeks after baseline)
  The MPQ is scored by summing the values of words that best describe a person's pain. The score ranges from 0 (no pain) to 78 (severe pain)
Change in Visual Analog Scale (VAS) to assess Pain | At baseline and at discharge (approximately 2-3 weeks after baseline)
  The VAS pain scale is a tool for assessing pain intensity. Participants will be asked to mark a point on a 100 mm horizontal line that represents the intensity of their pain. This line has two endpoints: 0: No pain and 100: Worst possible pain imaginable. The distance from the "0" to the mark is measured in millimeters with the resulting number (0-100) being the VAS pain score

CONTACTS AND LOCATIONS:
Overall Officials: Necolle Morgado-Vega, Principal Investigator — Yale University
Locations (1):
- Rehabilitation and Wellness Center at the Milford Campus of Bridgeport Hospital, Milford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No